CLINICAL TRIAL: NCT04069689
Title: A Phase I, Placebo-Controlled, Double-Blind, 2-Period Study to Assess Safety and Pharmacokinetics of Escalating Single and Multiple Oral Doses of EPX-100 in Fasting Healthy Subjects and Following a High-Fat Meal
Brief Title: Study of Safety and Pharmacokinetics of Oral Doses of EPX-100 in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Epygenix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EPX-100-002
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Dravet Syndrome
Keywords: Clemizole
MeSH Terms: conditions — Epilepsies, Myoclonic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- EPX-100 (Experimental): Single and multiple doses of 20, 40, 80mg of EPX-100 (Clemizole Hydrochloride)
  Interventions: Drug: EPX-100 (Clemizole Hydrochloride)
- Placebo (Placebo Comparator): Single and multiple doses of 20, 40, 80mg of placebo
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: EPX-100 (Clemizole Hydrochloride) — EPX-100 (Clemizole Hydrochloride)
  Other Names: Clemizole Hydrochloride; Clemizole HCL
  Arms: EPX-100
Drug: Placebos — Placebo to match EPX-100
  Arms: Placebo

SUMMARY:
This is a placebo-controlled, double-blind, 2-period study in 3 sequential groups of 8 healthy subjects each. The safety and pharmacokinetics of escalating single and multiple oral doses of EPX-100 will be assessed in fasting healthy subjects and following a high-fat meal.

DETAILED DESCRIPTION:
This is a placebo-controlled, double-blind, 2-period study in 3 sequential groups of 8 healthy subjects each. Subjects will be admitted on two occasions to the clinical research center: Day -1 for 14 days and discharged on Day 13 and then re-admitted on Day 19 for 3 days and discharged on Day 21. Subjects will fast after midnight on the day of each admission.

On Day 1 of study of the low-dose group (cohort 1), subjects will be randomized to a single dose of 20 mg EPX-100 (N=6) or placebo (N=2) in the morning and then remain fasting for 4 hours after dosing. Safety will be assessed and blood samples will be obtained to calculate PK at the following time points: 0, 0.5, 1, 2, 4, 6, 8, 12, 18, and 24 hours following the first dose of EPX-100 or placebo. The subjects will remain in the study research center for daily 8 AM (± 2 hours) blood samples for 5 consecutive days (Days 3 - 7; one blood sample per day). On Days 8 - 11, subjects will be administered 20 mg EPX-100 or placebo twice daily (BID) at least one hour prior to the morning meal and at least 2 hours after the evening meal (approximately 12 hours apart). A single dose of 20 mg EPX-100 or placebo will be administered on Day 12 in the fasting state and subjects will remain fasting for 4 hours after dosing. Blood samples will be drawn at the following time points: 0, 0.5, 1, 2, 4, 6, 8, 12, 18, and 24 hours to determine multiple-dose PK. After a washout period of at least one week following the last dose of EPX-100 or placebo, subjects will return to the clinical research center on Day 19 and safety will be assessed. On Day 20, subjects will ingest a high-fat morning meal over 30 minutes; thereafter, the subject will receive a single dose of 20 mg EPX- 100 or placebo at 30 minutes after the start of the meal. Blood samples will be drawn at the following time points: 0, 0.5, 1, 2, 4, 6, 8, 12, 18, and 24 hours after the administration of study drug to determine the PK of EPX-100 in the fed state. Once the 20 mg dose level of EPX-100 is evaluated and the Safety Review Committee (SRC) determines it is safe to escalate to the next dose level, subsequent groups of 8 subjects each will be administered 40 mg (cohort 2) and 80 mg (cohort 3) (N=6 active drug, N=2 matching placebo) EPX-100 and follow the same study procedures as the low-dose group (cohort 1).

Throughout the study period, subjects will undergo cardiac assessments, safety assessments, and PK sampling.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to any study-related procedures
2. Male or female subjects 18 to 50 years of age inclusive
3. Subject's body mass index (BMI) is ≤ 30 kg/m2
4. Female subjects of childbearing potential must not be pregnant or lactating with a negative serum human chorionic gonadotropin (HCG) pregnancy test result at Screening, Day -1, or Day 19.
5. Female subjects of childbearing potential and male subjects must use an adequate method of contraception from Screening until completion of the study. Acceptable methods of contraception are barrier methods (male condom, female condom, diaphragm, cervical cap, spermicide, or intrauterine device [IUD]), surgical sterility (documented doctor's report of vasectomy, hysterectomy, and/or bilateral oophorectomy), oral hormonal contraceptives, hormonal IUD, and/or postmenopausal status (defined as at least 1 year without menses as demonstrated by medical history or subject report).
6. Subject is in good health as determined by vital signs, medical history, physical exam, and safety laboratory analyses at Screening and during the study.

Exclusion Criteria:

1. Subject has used an investigational product within 30 days prior to enrollment or during the study.
2. Subject has used prescription or non-prescription drugs (including vitamins, minerals, and herbal/plant-derived preparations) within 2 weeks of enrollment (excluding oral hormonal contraceptives, hormonal IUD, hormone replacement therapy, and acetaminophen) unless deemed acceptable by the Investigator in consultation with the Sponsor.
3. Subject has a positive drug and/or alcohol test at Screening, Day -1, or Day 19.
4. Subject has a history of drug or alcohol abuse within 2 years before Screening.
5. Subject is unable to abstain from ingesting alcohol, caffeine, grapefruit or grapefruit juice, pomelo or pomelo juice, or Seville oranges or Seville orange juice for 72 hours prior to dosing and throughout the dosing periods.
6. Concurrent use of substances, including drugs, known to interfere with EPX-100, including moderate or severe inducers or inhibitors of CYP3A4 and CYP2D6.
7. The subject has a clinically significant history of endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major diseases or malignancy.
8. Subject has evidence of any of the following cardiac conduction abnormalities:

   1. QTcF interval >430 msec for males and >450 msec for females
   2. PR interval ⩾ 200 msec
   3. Evidence of second- or third-degree atrioventricular block (AVB)
   4. Electrocardiographic evidence of complete left bundle branch block (LBBB), complete right bundle branch block (RBBB), or incomplete LBBB
   5. Intraventricular conduction delay with QRS duration >120 msec
   6. Heart rate <40 bpm
   7. Pathological Q waves (defined as >40 msec or depth >0.4-0.5 mV)
   8. Evidence of ventricular pre-excitation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-27 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) | 21 days
  To evaluate the safety of single and multiple escalating doses of oral EPX-100 in healthy subjects.
Serial ECGs - QTcF Interval | 21 days
  To evaluate the safety of single and multiple escalating doses of oral EPX-100 in healthy subjects.
Physical Examinations Including Actual Body Weight | 21 days
  To evaluate the safety of single and multiple escalating doses of oral EPX-100 in healthy subjects.

SECONDARY OUTCOMES:
Plasma Concentrations of EPX-100 in Fasting State | 13 days
  Determine the pharmacokinetic (PK) profile of single and multiples doses of 20 mg, 40 mg, and 80 mg twice daily of EPX-100.
Plasma Concentration of EPX-100 following a High-Fat Meal | 24 hours
  Determine the PK profile of a single dose of EPX-100 in the fasting state compared with after a high-fat meal.

CONTACTS AND LOCATIONS:
Overall Officials: Hahn-Jun Lee, Ph.D., Study Director — Epygenix Therapeutics, Inc.
Locations (1):
- TKL Research, Fair Lawn, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No